CLINICAL TRIAL: NCT00534612
Title: Accuracy of Fine Needle Aspiration Biopsy in the Pre-Operative Diagnosis of Malignancy in Patients With Parotid Gland Masses
Brief Title: Diagnostic Accuracy of Fine Needle Aspiration in Parotid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 006/038/CCI
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2003-01

CONDITIONS: Parotid Gland Neoplasms
Keywords: Parotid gland neoplasms
MeSH Terms: interventions — Biopsy, Needle

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): fine needle aspiration biopsy of the parotid gland mass
  Interventions: Procedure: aspiration biopsy

INTERVENTIONS:
Procedure: aspiration biopsy — fine needle aspiration biopsy of the parotid gland masses

SUMMARY:
Liberal use of fine needle aspiration biopsy of parotid gland masses is controversial. All information regarding this procedure has been retrospective. Our objective is to evaluate prospectively the diagnostic accuracy of the test, alone and when associated to clinical and/or radiologic data.

DETAILED DESCRIPTION:
This is a prospective diagnostic test study. Inclusion criteria are all consecutive patients with parotid gland masses referred for treatment at our center, from January 2003 to December 2007.

The gold standard for the diagnosis of malignancy is the surgical pathology report of the parotidectomy specimen.

Cytologist and pathologist will be blind. Diagnostic accuracy is determinded by Bayesian analysis.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with parotid gland masses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of malignancy | three years

SECONDARY OUTCOMES:
Specific histopathologic diagnosis | three years

CONTACTS AND LOCATIONS:
Overall Officials: Jose F Carrillo, M.D:, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- National Cancer Institute, México, D.F:, Mexico